CLINICAL TRIAL: NCT02147821
Title: Necessity of Using Pleural Drainage Tubes After IMA Harvesting During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Aaron Spooner, MD, MMgt, HBSc, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: REB13-1374
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Pleural Effusions Post Coronary Artery Bypass Graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): Standard treatment will be defined as current practice whereby two mediastinal chest tubes are used for drainage, as well as an additional pleural tube if the pleura is opened during surgery. As part of current standard practice, the pleural and mediastinal spaces will be suctioned during the achievement of hemostasis prior to the insertion of chest tubes.
- Intervention (Experimental): The treatment arm of the study will involve standard placement of the mediastinal tubes with the exclusion of the pleural tube.
  Interventions: Procedure: No Pleural Chest Tube

INTERVENTIONS:
Procedure: No Pleural Chest Tube
  Arms: Intervention

SUMMARY:
This prospective randomized controlled trial will examine the efficacy of reducing the number of chest tubes used in the postoperative cardiac surgery patient. Typically used are three chest tubes - two in the mediastinum and one in the pleural space, if opened. The investigators propose that removal of the pleural tube will not impact the rates of clinically significant pleural effusions post cardiac surgery. Patients will be randomized into two groups - one receiving the standard three chest tubes (standard), and the other receiving only mediastinal drains (experimental). The primary outcome will be rates of post-operative pleural effusions as determined by defined interventions, including insertion of a chest tube, thoracentesis, or return to the operating room for primary evacuation of pleural effusion or hemothorax. Secondary outcomes include length of hospital stay, length of mechanical ventilation, postoperative respiratory status, and presence/size of pleural effusions, as well as readmission for pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* patients must be undergoing CABG at our institution with the attempted harvest of a LIMA and/or RIMA
* pleura must be entered in order for patients to be included.

Exclusion Criteria:

* cardiac surgery where the pleura is not entered
* previous surgery where the pleura was entered
* other pre-existing pleural diseases or fibrosis
* Patients currently participating in other studies
* Patients presenting with emergent need for bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-08; Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pleural Effusion | 6 weeks
  Primary outcome is rate of pleural effusions in a 6 week postoperative period of CABG.

SECONDARY OUTCOMES:
Postoperative Respiratory Status | 1 week after CABG
  Respiratory status will be defined by measurement of oxygen requirement as well as documented levels of incentive spirometry, as well as length of mechanical ventilation in ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada